CLINICAL TRIAL: NCT03987646
Title: The Vestibular Socket Therapy : A Novel Concept for Immediate Implant Placement in Defective Fresh Extraction Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nonstaged socket therapy
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Immediate Implants
Keywords: xenograft cortical flexible sheet; fresh extraction socket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- xenograft cortical flexible sheet (Experimental): a-traumatic tooth removal , socket lavage and curettage, performing a vestibular access horizontal incision corresponding to the socket 3-4 mm apically from the muccogingival junction , a tunnel is then created from the socket office and extended apically till it connects with the vestibular access incision, a computer guided surgical template is then used to deliver the implant in its optimal position, a slowly resorbable membrane shield is then introduced through the tunnel and stabilized with a membrane tac , it is a sturdy fixable membrane barrier placed above the labial plate
  Interventions: Procedure: Non-staged vestibular fresh socket therapy

INTERVENTIONS:
Procedure: Non-staged vestibular fresh socket therapy — a slowly resorbable membrane shield is placed above the labial plate of bone so that when the thin labial plate started its resorption process the shield remains till a complete gap fill occurred thus leading to a thicker labial plate of bone or it preserves the socket architecture until a complete bone fill occurred inside the socket
  Other Names: osteoflex

SUMMARY:
This article aims to provide a non- staged treatment protocol to placing dental implants in compromised fresh sockets in the aesthetic zone.

DETAILED DESCRIPTION:
This is a site-specific therapy uses study a slowly resorbing regenerative barrier (shield) to augment any thin or deficient labial plate of bone, enhances the overlying soft tissue quality and quantity at the same time with implant fixture placement using a computer-guided surgical template.

ELIGIBILITY:
Inclusion Criteria:

* A hopeless single tooth in the maxillary anterior region
* Sufficient apical bone to allow adequate anchorage/primary stability of the implant
* had natural teeth present adjacent to the tooth being replaced

Exclusion Criteria:

* Presence of acute infection
* Impossibility of reaching adequate implant primary stability in the native
* Smokers of > 10 cigarettes
* Antitumor chemotherapy or radiotherapy in the previous year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
radiographic buccal bone thickness | 6 months
  preoperative and follow up CBCTs are superimposed on each other and buccal bone thickness is measure at 3 similar points on both CBCTs and then a mean is calculated
radiographic buccal bone height | 6 months
  preoperative and follow up CBCTs are superimposed on each other and buccal bone height is measured in relation to implant shoulder level

SECONDARY OUTCOMES:
final esthetic outcome of soft tissue | 6 months
  Pink esthetic score. based on subjective assessment of mesial papilla, distal papilla, midfacial level, midfacial contour, alveolar process deficiency, soft tissue color and texture. each item is given a score between 0 and 2, where 0 is the worst and 2 is the best outcome. Then, a final score ranging between 0-14 is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Abdelsalam Elaskary, Study Chair — University of New York; Yasmine Y Gaweesh, PhD, Principal Investigator — Alexandria University; Paul Rosen, DMD, Principal Investigator — University of Maryland Dental School, Baltimore; Moataz Meabed, Msc, Principal Investigator — Oral Medicine and Periodontology, Cairo University. Egypt; Sang-Choon Cho, DDS, Study Director — NYU College of Dentistry, USA.
Locations (1):
- Private Practice Clinic, Alexandria, Egypt

REFERENCES:
- [Background] Chen ST, Buser D. Esthetic outcomes following immediate and early implant placement in the anterior maxilla--a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:186-215. doi: 10.11607/jomi.2014suppl.g3.3. PMID 24660198
- [Background] Chen ST, Buser D. Clinical and esthetic outcomes of implants placed in postextraction sites. Int J Oral Maxillofac Implants. 2009;24 Suppl:186-217. PMID 19885446
- [Background] Meijer HJA, Slagter KW, Vissink A, Raghoebar GM. Buccal bone thickness at dental implants in the maxillary anterior region with large bony defects at time of immediate implant placement: A 1-year cohort study. Clin Implant Dent Relat Res. 2019 Feb;21(1):73-79. doi: 10.1111/cid.12701. Epub 2018 Dec 11. PMID 30548160
- [Background] Barroso-Panella A, Gargallo-Albiol J, Hernandez-Alfaro F. Evaluation of Bone Stability and Esthetic Results After Immediate Implant Placement Using a Novel Synthetic Bone Substitute in the Anterior Zone: Results After 12 Months. Int J Periodontics Restorative Dent. 2018 Mar/Apr;38(2):235-243. doi: 10.11607/prd.2863. PMID 29447317